CLINICAL TRIAL: NCT04908982
Title: Aspirin for the Prevention of Preeclampsia in Women With Stage 1 Hypertension: A Pilot Study
Brief Title: Aspirin for the Prevention of Preeclampsia in Women With Stage 1 Hypertension
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eastern Virginia Medical School (Other)
Collaborators: AMAG Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: AS1H
Record Dates: First submitted 2021-05-26; First posted 2021-06-01 (Actual); Last update posted 2021-06-28 (Actual); Status verified 2021-05

CONDITIONS: Pre-Eclampsia
Keywords: Preeclampsia; Hypertension; Stage 1 Hypertension; Pregnancy; Aspirin; Low Dose Aspirin
MeSH Terms: conditions — Pre-Eclampsia; Hypertension | interventions — Aspirin

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to either receive 81mg of aspirin daily beginning between 12 and 16 weeks of pregnancy or to receive no aspirin.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: The Principal Investigator, Co-Investigators, and Sonographers will all be masked from knowledge of the intervention assigned to each participant. Participants and the Study Coordinator will not be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Aspirin (Experimental): Participants in this arm will be instructed to take 1 81mg aspirin daily beginning between weeks 12 and 16 of pregnancy and continuing until delivery.
  Interventions: Drug: Aspirin 81mg
- No Aspirin (No Intervention): Participants in this arm will receive no aspirin.

INTERVENTIONS:
Drug: Aspirin 81mg — 81mg aspirin daily beginning between 12 and 16 weeks of pregnancy and continuing until delivery.
  Arms: Aspirin

SUMMARY:
In 2017, the American College of Cardiology and the American Heart Association changed the diagnostic criteria for hypertension in non-pregnant adults. The parameters for the diagnosis of stage 1 hypertension were revised from a systolic blood pressure (BP) of 140 to 130 mm Hg and a diastolic BP of 90 to 80 mm Hg. Based on new criteria, stage 1 hypertension is associated with a 2-3 fold increased risk of preeclampsia. There are no data regarding prevention of preeclampsia in women with stage 1 hypertension. Low-dose aspirin has been used during pregnancy to prevent preeclampsia for women at high-risk for preeclampsia. Although the precise mechanism remains uncertain, it is possible that low-dose aspirin improves placental perfusion, which results in a decreased rate of preeclampsia. A study that examines the effect of low-dose aspirin on placenta vasculature and tissue elastography by using novel ultrasound tools would be useful. The 2017 Aspirin for Evidence-Based Preeclampsia Prevention trial compared 150 mg aspirin with placebo in women at high-risk of preeclampsia based on a first-trimester screening. They found a significant decrease in the rate of preterm preeclampsia (4.3% vs. 1.6%; P <0.01). Since this study used the screening algorithm including first-trimester serum markers and uterine artery Doppler, the generalizability in the U.S. women with stage 1 hypertension is limited. Our pilot study will examine 1) the effect of low-dose aspirin 81 mg in women with stage 1 hypertension on placental vasculature and shear-wave elastography; 2) the rate of preterm preeclampsia in women with stage 1 hypertension in a control group and in pregnancies treated with low-dose aspirin 81 mg; 3) feasibility of conducting a larger multicenter randomized controlled trial on this subject.

DETAILED DESCRIPTION:
In 2017, the American College of Cardiology (ACC) and the American Heart Association (AHA) changed the diagnostic criteria for hypertension in non-pregnant adults.1 The parameters for the diagnosis of stage 1 hypertension were revised from a systolic blood pressure (BP) of 140 to 130 mm Hg and a diastolic BP of 90 to 80 mm Hg.2 Stage 1 hypertension based on the new criteria is associated with an increased risk of preeclampsia compared to normal BP (15-16% vs. 5-7%).3, 4 However, the American College of Obstetricians and Gynecologists (ACOG) continues to diagnose chronic hypertension in pregnancy as a systolic BP above 140 mm Hg and a diastolic BP of 90 mm Hg since there are no data regarding prevention of preeclampsia in women with stage 1 hypertension.5

Preeclampsia is a multi-organ, progressive disorder characterized by the new onset of hypertension with proteinuria or end-organ dysfunction.6 Preeclampsia is a major cause of morbidity such as eclampsia, pulmonary edema, myocardial infarction, stroke, coagulopathy, and renal failure and a leading cause of iatrogenic preterm birth and maternal mortality.7 Preeclampsia is also an economic burden to the health care system. The mean combined maternal and infant medical care costs for women with preeclampsia are significantly higher than those of uncomplicated women ($41,790 vs. $13,187 in 2015 dollars) with the main cost drivers being infant health care costs due to prematurity.8

It is hypothesized that preeclampsia is caused by an imbalance in prostacyclin and thromboxane A2 (TXA2) resulting in vascular disturbances and coagulation defects. Low-dose aspirin (60-150 mg/day) irreversibly acetylates cyclooxygenase (COX)-1, which results in decreased platelet synthesis of TXA2 without affecting vascular wall production of prostacyclin.9. 10 However, it is likely that preeclampsia is a result of poor placentation. In this pilot study, we will examine the effect of low-dose aspirin on placental perfusion by using novel ultrasound tools (Superb Micro-Vascular Imaging [SMI], Shear Wave Elastography [SWE], intensity analysis [IA], and Attenuation Imaging [ATI]). Superb Micro-Vascular Imaging (SMI) is a novel Doppler technique designed to improve the visualization of microscopic vessels, through a new adaptive algorithm, which dramatically enhances microvascular flow and removes artifacts. Shear Wave Elastography (SWE) is a new noninvasive ultrasound-based technology for the evaluation of soft tissue stiffness. Intensity Analysis (IA) is a technique that analyzes tissue homogeneity. Attenuation Imagining (ATI) measures beam attenuation by quantifying an attenuation coefficient (AC db/cm/MHz). Our group has developed longitudinal nomograms on placental vasculature to include uterine and spiral arteries on the maternal side and fetal placental arterioles and umbilical artery on the fetal side.11 Furthermore, longitudinal nomograms related to placental tissue structure, including shear wave elastography has been developed.12

Although the precise mechanism is uncertain, low-dose aspirin has been used during pregnancy to prevent or delay the onset of preeclampsia for women at high-risk for preeclampsia.13 The 2017 Aspirin for Evidence-Based Preeclampsia Prevention trial compared 150 mg aspirin with placebo in women at high-risk of preeclampsia based on a first-trimester screening.14 They found a significant decrease in the rate of preterm preeclampsia less than 37 weeks of gestation (4.3% vs. 1.6%; P <0.01). Since this study used the screening algorithm including first-trimester serum markers and uterine artery Doppler, the generalizability of aspirin preeclampsia prevention in the U.S. women with stage 1 hypertension is limited.

Our long-term goal is to reduce preterm preeclampsia in women with stage 1 hypertension. We hypothesize that 1) spiral artery Pulsatility Index (PI) and Peak Systolic Velocity (PSV) and SWE is lower in women with stage 1 hypertension who receive low-dose aspirin 81 mg compared to those who do not receive low-dose aspirin; 2) Women with stage 1 hypertension who receive low-dose aspirin 81 mg have a lower rate of preterm preeclampsia compared to those who do not receive low-dose aspirin. To examine these hypotheses in a future, large randomized, controlled trial, our aims for this pilot study include the following:

Aim 1. To examine the change in placental vasculature and tissue elastography in women with stage 1 hypertension who receive low-dose aspirin 81 mg and those who do not receive low-dose aspirin.

Aim 2. To examine rates of preterm preeclampsia in women with stage 1 hypertension who receive low-dose aspirin 81 mg and those who do not receive low-dose aspirin.

Aim 3. To examine eligibility rate, recruitment rate, study compliance, and loss of follow-up rate. This information will be useful to assess feasibility of a future multicenter randomized controlled trial.

In summary, women with stage 1 hypertension are at an increased risk of preeclampsia. Low-dose aspirin may reduce the rate of preterm preeclampsia in women with stage 1 hypertension. In this pilot study, we will conduct an open label randomized controlled trial and obtain necessary information for a future multicenter randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women from 6 0/7 to 13 6/7 weeks gestation
* 18-50 years old
* Systolic blood pressure of 130-139 mmHg or Diastolic blood pressure of 80-89 mmHg

Exclusion Criteria:

* History of preeclampsia
* Multifetal gestation
* Chronic hypertension
* Pre-gestational diabetes
* Renal disease
* Autoimmune disease
* Aspirin allergy or hypersensitivity
* Presence of nasal polyps
* History of aspirin-induced bronchospasm

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-05-28 (Actual); Primary Completion 2023-05-31 (Estimated); Study Completion 2023-05-31 (Estimated)

PRIMARY OUTCOMES:
Preterm Preeclampsia | Prior to 37 weeks
  Preeclampsia developed before 37 weeks

SECONDARY OUTCOMES:
Preeclampsia | After 37 weeks
  Systolic blood pressure of 140 mmHg or more or diastolic blood pressure of 90 mmHg or more on two occasions at least four hours apart or a systolic blood pressure of 160 mmHg or more or diastolic blood pressure of 110 mmHg or more; and Proteinuria of 300mg or more per 24-hour urine collection or protein/creatinine ratio of 0.3 or more; or in the absence of proteinuria, new-onset hypertension with the new onset of any of the following severe features: thrombocytopenia, renal insufficiency, impaired liver function, pulmonary edema, new-onset headache unresponsive to medication.
Gestational Hypertension | After 20 weeks gestation
  Systolic blood pressure of 140 mmHg or more or diastolic blood pressure of 90 mmHg or more on two occasions at least four hours apart with no proteinuria or severe features.
HELLP Syndrome | After 20 weeks gestation
  Hemolysis, elevated liver enzymes, and low platelet count syndrome
Eclampsia | After 20 weeks gestation
  New-onset tonic-clonic, focal, or multifocal seizure in the absence of other causative conditions

CONTACTS AND LOCATIONS:
Overall Officials: Tetsuya Kawakita, MD, Principal Investigator — Eastern Virginia Medical School
Locations (1):
- Department of Obstetrics and Gynecology, Division of Maternal-Fetal Medicine, Eastern Virginia Medical School, Norfolk, Virginia, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Whelton PK, Carey RM, Aronow WS, Casey DE Jr, Collins KJ, Dennison Himmelfarb C, DePalma SM, Gidding S, Jamerson KA, Jones DW, MacLaughlin EJ, Muntner P, Ovbiagele B, Smith SC Jr, Spencer CC, Stafford RS, Taler SJ, Thomas RJ, Williams KA Sr, Williamson JD, Wright JT Jr. 2017 ACC/AHA/AAPA/ABC/ACPM/AGS/APhA/ASH/ASPC/NMA/PCNA Guideline for the Prevention, Detection, Evaluation, and Management of High Blood Pressure in Adults: Executive Summary: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines. Hypertension. 2018 Jun;71(6):1269-1324. doi: 10.1161/HYP.0000000000000066. Epub 2017 Nov 13. No abstract available. PMID 29133354
- [Background] Topel ML, Duncan EM, Krishna I, Badell ML, Vaccarino V, Quyyumi AA. Estimated Impact of the 2017 American College of Cardiology/American Heart Association Blood Pressure Guidelines on Reproductive-Aged Women. Hypertension. 2018 Oct;72(4):e39-e42. doi: 10.1161/HYPERTENSIONAHA.118.11660. PMID 30354726
- [Background] Hauspurg A, Parry S, Mercer BM, Grobman W, Hatfield T, Silver RM, Parker CB, Haas DM, Iams JD, Saade GR, Wapner RJ, Reddy UM, Simhan H. Blood pressure trajectory and category and risk of hypertensive disorders of pregnancy in nulliparous women. Am J Obstet Gynecol. 2019 Sep;221(3):277.e1-277.e8. doi: 10.1016/j.ajog.2019.06.031. Epub 2019 Jun 27. PMID 31255629
- [Background] Sutton EF, Hauspurg A, Caritis SN, Powers RW, Catov JM. Maternal Outcomes Associated With Lower Range Stage 1 Hypertension. Obstet Gynecol. 2018 Oct;132(4):843-849. doi: 10.1097/AOG.0000000000002870. PMID 30204698
- [Background] Battarbee AN, Sinkey RG, Harper LM, Oparil S, Tita ATN. Chronic hypertension in pregnancy. Am J Obstet Gynecol. 2020 Jun;222(6):532-541. doi: 10.1016/j.ajog.2019.11.1243. Epub 2019 Nov 9. PMID 31715148
- [Background] Steegers EA, von Dadelszen P, Duvekot JJ, Pijnenborg R. Pre-eclampsia. Lancet. 2010 Aug 21;376(9741):631-44. doi: 10.1016/S0140-6736(10)60279-6. Epub 2010 Jul 2. PMID 20598363
- [Background] ACOG Practice Bulletin No. 202: Gestational Hypertension and Preeclampsia. Obstet Gynecol. 2019 Jan;133(1):1. doi: 10.1097/AOG.0000000000003018. PMID 30575675
- [Background] Hao J, Hassen D, Hao Q, Graham J, Paglia MJ, Brown J, Cooper M, Schlieder V, Snyder SR. Maternal and Infant Health Care Costs Related to Preeclampsia. Obstet Gynecol. 2019 Dec;134(6):1227-1233. doi: 10.1097/AOG.0000000000003581. PMID 31764733
- [Background] Clarke RJ, Mayo G, Price P, FitzGerald GA. Suppression of thromboxane A2 but not of systemic prostacyclin by controlled-release aspirin. N Engl J Med. 1991 Oct 17;325(16):1137-41. doi: 10.1056/NEJM199110173251605. PMID 1891022
- [Background] Patrono C. Aspirin as an antiplatelet drug. N Engl J Med. 1994 May 5;330(18):1287-94. doi: 10.1056/NEJM199405053301808. No abstract available. PMID 8145785
- [Background] Horgan R, Sinkovskaya E, Saade G, Kalafat E, Rice MM, Heeze A, Abuhamad A. Longitudinal assessment of spiral and uterine arteries in normal pregnancy using novel ultrasound tool. Ultrasound Obstet Gynecol. 2023 Dec;62(6):860-866. doi: 10.1002/uog.26312. PMID 37470712
- [Background] Abuhamad A, Sinkovskaya E, Heeze A, et al. Longitudinal assessment of placental shear-wave elastography and correlation with placental circulation in normal pregnancies. Am J Obstet Gynecol. 2020;222(1)S67
- [Background] ACOG Committee Opinion No. 743: Low-Dose Aspirin Use During Pregnancy. Obstet Gynecol. 2018 Jul;132(1):e44-e52. doi: 10.1097/AOG.0000000000002708. PMID 29939940
- [Background] Rolnik DL, Wright D, Poon LC, O'Gorman N, Syngelaki A, de Paco Matallana C, Akolekar R, Cicero S, Janga D, Singh M, Molina FS, Persico N, Jani JC, Plasencia W, Papaioannou G, Tenenbaum-Gavish K, Meiri H, Gizurarson S, Maclagan K, Nicolaides KH. Aspirin versus Placebo in Pregnancies at High Risk for Preterm Preeclampsia. N Engl J Med. 2017 Aug 17;377(7):613-622. doi: 10.1056/NEJMoa1704559. Epub 2017 Jun 28. PMID 28657417
- [Background] Muntner P, Carey RM, Gidding S, Jones DW, Taler SJ, Wright JT Jr, Whelton PK. Potential US Population Impact of the 2017 ACC/AHA High Blood Pressure Guideline. Circulation. 2018 Jan 9;137(2):109-118. doi: 10.1161/CIRCULATIONAHA.117.032582. Epub 2017 Nov 13. PMID 29133599
- [Background] Duley L, Henderson-Smart DJ, Meher S, King JF. Antiplatelet agents for preventing pre-eclampsia and its complications. Cochrane Database Syst Rev. 2007 Apr 18;(2):CD004659. doi: 10.1002/14651858.CD004659.pub2. PMID 17443552
- [Background] Askie LM, Duley L, Henderson-Smart DJ, Stewart LA; PARIS Collaborative Group. Antiplatelet agents for prevention of pre-eclampsia: a meta-analysis of individual patient data. Lancet. 2007 May 26;369(9575):1791-1798. doi: 10.1016/S0140-6736(07)60712-0. PMID 17512048
- [Background] Henderson JT, Whitlock EP, O'Connor E, Senger CA, Thompson JH, Rowland MG. Low-dose aspirin for prevention of morbidity and mortality from preeclampsia: a systematic evidence review for the U.S. Preventive Services Task Force. Ann Intern Med. 2014 May 20;160(10):695-703. doi: 10.7326/M13-2844. PMID 24711050
- [Background] CLASP: a randomised trial of low-dose aspirin for the prevention and treatment of pre-eclampsia among 9364 pregnant women. CLASP (Collaborative Low-dose Aspirin Study in Pregnancy) Collaborative Group. Lancet. 1994 Mar 12;343(8898):619-29. PMID 7906809
- [Background] Ahrens KA, Silver RM, Mumford SL, Sjaarda LA, Perkins NJ, Wactawski-Wende J, Galai N, Townsend JM, Lynch AM, Lesher LL, Faraggi D, Zarek S, Schisterman EF. Complications and Safety of Preconception Low-Dose Aspirin Among Women With Prior Pregnancy Losses. Obstet Gynecol. 2016 Apr;127(4):689-698. doi: 10.1097/AOG.0000000000001301. PMID 26959198
- [Background] Slone D, Siskind V, Heinonen OP, Monson RR, Kaufman DW, Shapiro S. Aspirin and congenital malformations. Lancet. 1976 Jun 26;1(7974):1373-5. doi: 10.1016/s0140-6736(76)93025-7. PMID 59014
- [Background] Kozer E, Nikfar S, Costei A, Boskovic R, Nulman I, Koren G. Aspirin consumption during the first trimester of pregnancy and congenital anomalies: a meta-analysis. Am J Obstet Gynecol. 2002 Dec;187(6):1623-30. doi: 10.1067/mob.2002.127376. PMID 12501074
- [Background] Wyatt-Ashmead J. Antenatal closure of the ductus arteriosus and hydrops fetalis. Pediatr Dev Pathol. 2011 Nov-Dec;14(6):469-74. doi: 10.2350/07-11-0368.1. Epub 2011 Oct 10. PMID 21985268
- [Background] Pickering TG, Hall JE, Appel LJ, Falkner BE, Graves J, Hill MN, Jones DW, Kurtz T, Sheps SG, Roccella EJ. Recommendations for blood pressure measurement in humans and experimental animals: part 1: blood pressure measurement in humans: a statement for professionals from the Subcommittee of Professional and Public Education of the American Heart Association Council on High Blood Pressure Research. Circulation. 2005 Feb 8;111(5):697-716. doi: 10.1161/01.CIR.0000154900.76284.F6. PMID 15699287